CLINICAL TRIAL: NCT06591520
Title: A Randomized, Controlled, Multi-center Phase III Study of AK112 Combined With Gemcitabine Plus Cisplatin Versus Durvalumab Combined With Gemcitabine Plus Cisplatin as the First-line Treatment for Patients With Advanced Biliary Tract Cancer
Brief Title: AK112 Combined With Chemotherapy Versus Durvalumab Combined With Chemotherapy in Advanced Biliary Tract Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akeso (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK112-309
Record Dates: First submitted 2024-09-08; First posted 2024-09-19 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Gemcitabine; Cisplatin; durvalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AK112 + Gemcitabine + Cisplatin (Experimental)
  Interventions: Drug: AK112, Gemcitabine, Cisplatin
- Durvalumab + Gemcitabine + Cisplatin (Active Comparator)
  Interventions: Drug: Durvalumab, Gemcitabine, Cisplatin

INTERVENTIONS:
Drug: AK112, Gemcitabine, Cisplatin — AK112 will be administered at a selected dose intravenously (IV) every three weeks (Q3W). Gemcitabine will be administered at 1000 mg/m2, D1, D8, Q3W, intravenously (IV) for 8 cycles. Cisplatin will be administered at 25 mg/m2, D1, D8, Q3W, intravenously (IV) for 8 cycles.
  Arms: AK112 + Gemcitabine + Cisplatin
Drug: Durvalumab, Gemcitabine, Cisplatin — Durvalumab will be administered at 1500mg intravenously (IV) every three weeks (Q3W) for 8 cycles and followed by monotherapy every 4 weeks. Gemcitabine will be administered at 1000 mg/m2, D1, D8, Q3W, intravenously (IV) for 8 cycles. Cisplatin will be administered at 25 mg/m2, D1, D8, Q3W, intravenously (IV) for 8 cycles.
  Arms: Durvalumab + Gemcitabine + Cisplatin

SUMMARY:
This is a phase 3 study. All subjects are patients with unresectable locally advanced or metastatic biliary tract cancer (BTC), Eastern Cooperative Oncology Group (ECOG) performance status 0-1. The purpose of this study is to evaluate the efficacy and safety of AK112 in combination with chemotherapy versus durvalumab in combination with chemotherapy in patients with unresectable locally advanced or metastatic BTC.

ELIGIBILITY:
Inclusion Criteria:

* Be able and willing to provide written informed consent.
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Has a life expectancy of at least 3 months.
* Has a histologically or cytologically confirmed diagnosis of biliary tract cancer (BTC).
* Has no prior systemic anti-tumor therapy for unresectable locally advanced or metastatic BTC.
* Has measurable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
* Has adequate organ function.

Exclusion Criteria:

* Has other malignancies within 5 years prior to enrollment.
* Is currently participating in a study of an investigational agent or using an investigational device.
* Has known active central nervous system (CNS) metastases.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years.
* Has an active infection requiring systemic therapy.
* Has known active Hepatitis B or Hepatitis C.
* History of myocardial infarction, unstable angina, congestive heart failure within 12 months prior to enrollment.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study.
* Has received a live virus vaccine within 30 days of the planned first dose of study therapy.
* Has any concurrent medical condition that, in the opinion of the Investigator, would complicate or compromise compliance with the study or the well-being of the subject.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 682 (Actual)
Dates: Start 2024-10-20 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to approximately 2 years
  OS is the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from randomization to the first documented disease progression (per RECIST v1.1 criteria) assessed by investigators or death due to any cause, whichever occurs first.
Objective Response Rate (ORR) | Up to approximately 2 years
  ORR is the proportion of subjects with complete response(CR) or partial response(PR) , assessed by investigators based on RECIST v1.1.
Duration of Response (DoR) | Up to approximately 2 years
  The DoR was defined as the time from the date of first documented OR (confirmed CR or confirmed PR) until date of documented progression (PD) based on investigator assessments by using RECIST version 1.1 or death in absence of disease progression.
Disease Control Rate (DCR) | Up to approximately 2 years
  DCR is the proportion of subjects with complete response(CR) , partial response (PR) or stable disease (SD) , assessed by investigators based on RECIST v1.1.
Time to response (TTR) | Up to approximately 2 years
  TTR is defined as the time to response based on RECIST v1.1.
Adverse Events (AEs) | Up to approximately 2 years
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Wenting Li, MD, Study Director — Akeso
Locations (2):
- China (2):
  - Harbin Medical University Cancer Hospital, Harbin
  - Zhongshan Hospital, Fudan University, Shanghai